CLINICAL TRIAL: NCT00538928
Title: Extrapulmonary Interventional Ventilatory Support for Lung Protection in Severe Acute Respiratory Distress - a Prospective Randomized Multi Centre Study
Brief Title: Extrapulmonary Interventional Ventilatory Support in Severe Acute Respiratory Distress Syndrome (ARDS)
Acronym: Xtravent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Department of Anesthesia, University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KKS 4012-001-07
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2009-03

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: acute respiratory distress syndrome; extracorporeal lung support; hypoxia; hypercapnia; acute respiratory distress syndrome (ARDS)
MeSH Terms: conditions — Respiratory Distress Syndrome; Hypoxia; Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intervention: Implantation of the iLA - adaptation of the ventilation strategy, explantation of the iLA after corresponding improvement (see treatment plan for details) - weaning from the ventilation and extubation according to specified criteria.
  Interventions: Other: lung protective ventilation
- 2 (Active Comparator): no device: Ventilation strategy based on the concept of lung-protective ventilation without extracorporeal support, weaning from the ventilation and extubation according to specified criteria (see treatment plan for details).
  Interventions: Other: lung protective ventilation

INTERVENTIONS:
Other: lung protective ventilation — tidal volume 6 ml/kg ideal body weight

SUMMARY:
A prospective, randomized study will be performed investigating the effects of a pumpless extracorporeal interventional lung assist [iLA] on the implementation of a lung-protective ventilatory strategy in patients with acute respiratory distress syndrome [ARDS] with a PaO2/FiO2 ratio < 200. The duration of ventilation, intensive care and hospital stay and in-hospital mortality will be investigated.

DETAILED DESCRIPTION:
Evaluation group:

Implantation of the iLA - adaptation of the ventilation strategy, explantation of the iLA after corresponding improvement (see treatment plan for details) - weaning from the ventilation and extubation according to specified criteria.

Control group:

Ventilation strategy based on the concept of lung-protective ventilation without extracorporeal support, weaning from the ventilation and extubation according to specified criteria (see treatment plan for details).

ELIGIBILITY:
Inclusion Criteria:

* The trial subjects are patients aged 18 years or older who have developed severe ARDS. Following the American-European Consensus Conference on ARDS, severe ARDS is defined as an oxygenation index (PaO2/FIO2) < 200 mmHg. These parameters must be present for a duration of at least 2 hours.

Exclusion Criteria:

* age < 18 years
* decompensated heart insufficiency
* acute coronary syndrome
* severe chronic obstructive pulmonary disease
* advanced tumour conditions with life expectancy < 6 months
* chronic dialysis treatment
* lung transplant patients
* proven Heparin-induced thrombocytopenia (HIT)
* morbid obesity (BMI >) 40
* Child Class B and C cirrhosis of the liver, acute fulminant hepatic failure
* severe peripheral arterial occlusive disease (pAVK III - IV), absence of limb doppler pulse
* brain injury (GCS < 9 + CT pathology)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Ventilator free days within 28 days after enrollment | 28 days

SECONDARY OUTCOMES:
hospital mortality, organ-failure free days, pulmonary gas exchange | 28 days - 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bein, Professor Dr., Principal Investigator — University Hospital Regensburg; Steffen Weber-Carstens, Dr., Study Chair — Charite University Hospital Berlin; Thomas Staudinger, Prof, Study Chair — University Hospital Vienna, Austria; Sven Bercker, MD, Study Chair — University Hospital Leipzig, Germany; Ralph Müllenbach, MD PhD, Study Chair — University Hospital Würzburg, Germany; Rolf Dembinski, MD PhD, Study Chair — University Hospital Aachen, Germany
Locations (1):
- University Hospital Regensburg, Regensburg, Germany

REFERENCES:
- [Background] Bein T, Weber F, Philipp A, Prasser C, Pfeifer M, Schmid FX, Butz B, Birnbaum D, Taeger K, Schlitt HJ. A new pumpless extracorporeal interventional lung assist in critical hypoxemia/hypercapnia. Crit Care Med. 2006 May;34(5):1372-7. doi: 10.1097/01.CCM.0000215111.85483.BD. PMID 16540950
- [Derived] Bein T, Weber-Carstens S, Goldmann A, Muller T, Staudinger T, Brederlau J, Muellenbach R, Dembinski R, Graf BM, Wewalka M, Philipp A, Wernecke KD, Lubnow M, Slutsky AS. Lower tidal volume strategy ( approximately 3 ml/kg) combined with extracorporeal CO2 removal versus 'conventional' protective ventilation (6 ml/kg) in severe ARDS: the prospective randomized Xtravent-study. Intensive Care Med. 2013 May;39(5):847-56. doi: 10.1007/s00134-012-2787-6. Epub 2013 Jan 10. PMID 23306584